CLINICAL TRIAL: NCT02911285
Title: Glial Regulators for Treating Comorbid Posttraumatic Stress Disorder and Substance Use Disorders
Brief Title: NAC for Treating Comorbid PTSD and SUD
Acronym: DoD-NAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Institute for Translational Neuroscience (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00052757
Record Dates: First submitted 2016-09-01; First posted 2016-09-22 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Alcohol Use Disorder (AUD); Substance Use Disorder (SUD)
Keywords: Alcohol; PTSD; Trauma; Veteran; Substance; Drug; Post Traumatic Stress Disorder; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Substance-Related Disorders; Wounds and Injuries | interventions — Acetylcysteine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC/CBT (Experimental): Participants will receive N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) for 8 weeks.
  Interventions: Drug: N-acetylcysteine; Behavioral: Cognitive behavioral therapy
- Placebo/CBT (Placebo Comparator): Participants will receive placebo pills and CBT for 8 weeks.
  Interventions: Drug: Placebo; Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Drug: N-acetylcysteine — 1200mg bid (2400mg/day)
  Other Names: NAC
  Arms: NAC/CBT
Drug: Placebo — Placebo pills bid
  Arms: Placebo/CBT
Behavioral: Cognitive behavioral therapy — CBT for AUD/SUD, one hour/once a week
  Other Names: CBT

SUMMARY:
As a result of sustained operations in Afghanistan and Iraq, there are an increasing number of U.S. military Veterans with substance use disorders and comorbid posttraumatic stress disorder (PTSD). If left untreated, individuals with substance use disorders and PTSD are at increased risk for developing other mental health problems (e.g., depression, anxiety), suicidal ideation and attempts, medical problems, reduced resiliency and military readiness, vocational problems, and family/social impairment. This study will determine the benefits of N-acetylcysteine (NAC) in treating alcohol use disorder and comorbid post-traumatic stress disorder (PTSD) among military Veterans.

DETAILED DESCRIPTION:
As a result of sustained operations in Afghanistan and Iraq, there are an increasing number of U.S. military Veterans with substance use disorders and comorbid posttraumatic stress disorder (PTSD). While mental health services are in place for U.S. service members, substantial gaps in the treatment of co-occurring substance use disorders and PTSD exist and there is little scientific evidence available to guide the provision of care. Treatment for comorbid substance use disorders and PTSD, especially pharmacologic treatment, is largely ineffective and short-lived. While there have been numerous studies focused largely on dopaminergic mechanisms of reward, they have not led to the development of adequate treatments for comorbid substance use disorders and PTSD. Animal models demonstrate that (a) acute stress and chronic use of addictive substances reduce the capacity of glia to remove the neurotransmitter glutamate, and (b) this impairment as well as relapse can be prevented or reversed by N-acetylcysteine (NAC). Further, human studies indicate that NAC is associated with reduced craving and substance use. Based on this, the investigators conducted a Proof of Principle (PoP) study which was the first to examine the use of NAC for the treatment of PTSD, with or without comorbid addiction. In this randomized, controlled double-blind pilot study the investigators showed that Veterans with substance use disorders (81.5% alcohol use disorder) and PTSD who were treated with 2400mg NAC for 8 weeks demonstrated significant reduction in PTSD severity and craving. Moreover, reductions in PTSD and substance-related symptomatology were sustained at 1-month follow-up. However, to extend and confirm its clinical utility in the military/Veteran context, it is important to know whether NAC reduces severity of alcohol use disorder (AUD), the most common addiction among Veterans and military service members, and the mechanisms underlying therapeutic response. Based on promising data from the PoP project, the proposed Extend-and-Confirm (EC) study will determine the efficacy of NAC in reducing AUD and comorbid PTSD in Veterans (N=90). Further, new aims include the application of functional magnetic resonance imaging (fMRI) and proton magnetic resonance spectroscopy (1H-MRS) to investigate the pathophysiology of AUD/PTSD, as well as prognostic indicators of treatment outcome. These aims extend the Future Plans proposed in the original PoP study and provide an opportunity for collaboration among clinical and preclinical investigators at the Ralph H. Johnson Veterans Affairs (VA) Medical Center and the Medical University of South Carolina (MUSC) to solve this critical health problem in the military context. In the proposed EC study, the investigators will (1) employ a randomized, double-blind, between-groups experimental design that will consist of 8 weeks of treatment with NAC (2400mg) or placebo medication, and follow-up assessment at 1-, 3-, and 6-months post treatment; (2) use standardized, repeated dependent measures to rigorously assess AUD severity and PTSD symptomatology during treatment and follow-up; (3) collect biologic measures of alcohol use; (4) measure impairment in associated areas of functioning (e.g., depression, sleep, suicidality, risky sexual behaviors, family/social functioning); and (5) employ advanced neuroimaging techniques before and after treatment among a subset of enrolled subjects. This proposal is directly responsive to the missions of the Institute for Translational Neuroscience (ITN), and the US Army/Department of Defense (DoD) in that it seeks to accelerate the development of new, medication-based treatments to mitigate the impact of AUD and comorbid psychological conditions, such as PTSD, in the military/Veteran context. The findings of this study will provide critically needed empirical evidence to help inform practice guidelines and better serve the needs of U.S. service members, Veterans and their families.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any race or ethnicity, age 18 to 75 years old.
* U.S. military Veteran, including National Guard and Reservists.
* Able to comprehend English.
* Meet Diagnostic and Statistical Manual (DSM-5) criteria for current alcohol use disorder (AUD) and/or substance use disorder (SUD).
* Meet DSM-5 criteria for current PTSD or subthreshold PTSD. Subjects may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or other anxiety disorders (e.g., panic disorder, agoraphobia, social phobia, generalized anxiety disorder). The inclusion of subjects with affective and other anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with PTSD (Brady et al., 2000; Kessler et al., 2005).
* Subjects taking psychotropic medications will be required to be maintained on a stable dose for at least four weeks before treatment initiation. This is because initiation or change of medications during the course of the trial may interfere with interpretation of results.
* Must consent to random assignment to N-acetylcysteine (NAC) or placebo.
* Must consent to complete all treatment and follow-up visits.

Exclusion Criteria:

* Subjects meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders, as the study protocol may be therapeutically insufficient.
* Subjects with a current eating disorder (bulimia, anorexia nervosa) or with dissociative identity disorder, as they are likely to require specific time-intensive psychotherapy.
* Subjects experiencing significant withdrawal symptoms, as evidence by a score of 10 or above on the Clinical Institute Withdrawal Assessment of Alcohol (CIWA).These subjects will be referred for clinical detoxification and may be re-assessed for study eligibility after medically supervised detoxification has been completed.
* Individuals considered an immediate suicide risk based on the Columbia Suicide Severity Rating Scale (C-SSRS) or who are likely to require hospitalization during the course of the study.
* Women who are pregnant, nursing or not practicing an effective form of birth control.
* Asthma or any clinically significant medical condition that in the opinion of the investigators would adversely affect safety or study participation.
* Use of carbamazepine, phenytoin, nitrous oxide, methotrexate, 6 azauridine triacetate, or nitroglycerin within the last 14 days or any other medication felt to have a hazardous interaction if taken with NAC.
* History of childhood or adult seizures of any cause.
* MRI exclusions: Claustrophobia; tattoos above the shoulders; permanent eyeliner or permanent artificial eyebrows; cardiac pacemaker; metal fragments in eye, skin, or body, including shrapnel; heart valve replacement; brain clips; venous umbrella; being a sheet-metal worker or welder; lifetime history of aneurysm surgery; intracranial bypass, renal, or aortic clips; prosthetic devices such as middle ear, eye, joint, or penile implants; joint replacements; non-removable hearing aid, neurostimulator, or insulin pump; shunts/stents; metal mesh/coil implants; metal plate/pin/screws/wires; or any other metal implants. Note that individuals who meet inclusion/exclusion criteria for the medication component of the study but not the MRI portion (e.g., excluded due to metal implants) will still be eligible to enroll in and complete the medication/treatment phase.
* Subjects on maintenance anxiolytic, antidepressant, or mood stabilizing medications which have been initiated during the past four weeks. If it is determined, based on clinical criteria, that a subject needs to be started on maintenance medications for anxiety, mood or psychotic symptoms during the course of the study, they will be discontinued from the treatment trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudie Back, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetylcysteine (NAC) Plus Cognitive Behavioral Therapy (CBT): Participants randomized to N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) for 8 weeks.
  N-acetylcysteine: 1200mg bid (2400mg/day)
  Cognitive behavioral therapy: CBT for AUD/SUD, one hour/once a week
- Placebo + Cognitive Behavioral Therapy (CBT): Participants received placebo pills and Cognitive Behavioral Therapy (CBT) for 8 weeks.
  Placebo: Placebo pills bid
  Cognitive behavioral therapy: CBT for AUD/SUD, one hour/once a week
Period: Overall Study
Arm/Group | N-acetylcysteine (NAC) Plus Cognitive Behavioral Therapy (CBT) | Placebo + Cognitive Behavioral Therapy (CBT)
Started | 49 | 41
Completed | 40 | 36
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 8 | 5
Not completed — Participant got a job and no longer had time to participate. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- N-acetylcysteine + Cognitive Behavioral Therapy: Participants received N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) for 8 weeks.
  N-acetylcysteine: 1200mg bid (2400mg/day)
  Cognitive behavioral therapy: CBT for AUD/SUD, one hour/once a week
- Placebo + Cognitive Behavioral Therapy: Participants received placebo pills and CBT for 8 weeks.
  Placebo: Placebo pills bid
  Cognitive behavioral therapy: CBT for AUD/SUD, one hour/once a week
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine + Cognitive Behavioral Therapy | Placebo + Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 49 | 41 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.99 (11.51) | 49.13 (13.23) | 50.85 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants] — Data on sex collected via self-report demographic form.
  Participants
    Female | 5 | 2 | 7
    Male | 44 | 39 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 46 | 40 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 20 | 46
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 49 | 41 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use Disorder Severity
Description: Change in Alcohol Use Disorder Severity as measured by change in average drinking days per week from baseline to week 8.
  Greater reduction in drinking days indicates better treatment outcomes. Drinking days measured over 1 week periods (7 days). Scale ranges from 0 days to 7 days.
Time Frame: From baseline to week 8 of treatment
Measure: Mean (Standard Deviation); unit: drinking days reduction
Groups:
- N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT): Participants received N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) for 8 weeks.
  N-acetylcysteine: 1200mg twice per day (2400mg/day)
  Cognitive behavioral therapy: for alcohol/substance use disorder, one hour/once a week
- Placebo and Cognitive Behavioral Therapy (CBT): Participants received placebo pills and CBT for 8 weeks.
  Placebo: Placebo pills twice per day
  Cognitive behavioral therapy: for alcohol/substance use disorder, one hour/once a week
Arm/Group | N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) | Placebo and Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 40 | 36
drinking days reduction | -2.65 (3.85) | -2.82 (4.86)

2. Primary Outcome: Change in Post Traumatic Stress Disorder Severity
Description: Change in post traumatic stress disorder severity as measured by Change in Clinician Administered PTSD Scale (CAPS-5) score from baseline to week 8.
  Greater change/reduction in score indicates better outcomes and greater reduction in PTSD symptomatology.
  (minimum score of 0 = absent to a maximum score of 80 = extreme)
Time Frame: From baseline to week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT): Participants received N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) for 8 weeks.
  N-acetylcysteine: 1200mg bid (2400mg/day)
  Cognitive behavioral therapy: CBT for AUD/SUD, one hour/once a week
- Placebo and Cognitive Behavioral Therapy (CBT): Participants received placebo pills and CBT for 8 weeks.
  Placebo: Placebo pills bid
  Cognitive behavioral therapy: CBT for AUD/SUD, one hour/once a week
Arm/Group | N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) | Placebo and Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 40 | 36
score on a scale | -6.93 (13.42) | -5.53 (11.10)

3. Primary Outcome: Change in Alcohol Craving
Description: Change in Alcohol craving as measured by change in Obsessive Compulsive Drinking Scale (OCDS) Total Score.
  Greater change/reduction in score indicates better outcomes and reduced alcohol craving.
  (Scores range from 0 to 56)
Time Frame: From baseline to week 8
Population: 39 participants completed survey in NAC group and 37 participants completed survey in placebo group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) | Placebo and Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 39 | 37
score on a scale | -3.97 (7.26) | -2.92 (5.97)

4. Primary Outcome: Change in Post Traumatic Stress Disorder Severity
Description: Post traumatic stress disorder symptoms as measured by change/reduction in score of post traumatic stress disorder checklist (PCL-5) from baseline to week 8.
  Greater reduction in score indicates better treatment outcomes. (minimum score of 0 = absent to a maximum score of 80 = extreme)
Time Frame: From baseline to week 8
Population: 39 participants completed survey in NAC group, and 37 completed survey in placebo group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT): Participants received N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) for 8 weeks.
  N-acetylcysteine: 1200mg twice per day (2400mg/day)
  Cognitive behavioral therapy for alcohol/substance use disorder, one hour/once a week
- Placebo and Cognitive Behavioral Therapy (CBT): Participants received placebo pills and CBT for 8 weeks.
  Placebo: Placebo pills twice per day
  Cognitive behavioral therapy for alcohol/substance use disorder, one hour/once a week
Arm/Group | N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) | Placebo and Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 39 | 37
score on a scale | -12.97 (18.36) | -9.97 (16.75)

ADVERSE EVENTS:
Time Frame: Approximately 8-9 months.
Arm/Group | N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) | Placebo and Cognitive Behavioral Therapy (CBT)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/41
Serious Adverse Events (participants affected / at risk) | 3/49 | 2/41
Other Adverse Events (participants affected / at risk) | 30/49 | 28/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) (N=49) | Placebo and Cognitive Behavioral Therapy (CBT) (N=41)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Aborted Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Liver Lesions (Hepatobiliary disorders) | 0 (0) | 1 (1)
Severe Nose Bleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (NAC) and Cognitive Behavioral Therapy (CBT) (N=49) | Placebo and Cognitive Behavioral Therapy (CBT) (N=41)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Fatigue (General disorders) | 5 (5) | 4 (4)
Flatulence (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 14 (14) — General respiratory illness (cold, cough, flu, sinus infection, congestion)
Appetite Changes (Metabolism and nutrition disorders) | 1 (1) | 3 (3) — Increase or decrease in appetite
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT02911285/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT02911285/ICF_001.pdf